CLINICAL TRIAL: NCT03758352
Title: The Effect of Remote Ischemic Preconditioning on Ischemia/Reperfusion Injury in a Liver Transplant Recipient (TRSPLNT) - A Randomized, Controlled, Double-blinded Clinical Trial.
Brief Title: The Effect of Remote Ischemic Preconditioning on Ischemia/Reperfusion Injury in a Liver Transplant Recipient
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Large sample size
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Waqas Farooqui, MD, Principal Investigator, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TRSPLNT001
Record Dates: First submitted 2018-11-25; First posted 2018-11-29 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Liver Transplant; Complications; Ischemia Reperfusion Injury
Keywords: ischemia reperfusion injury; remote ischemic preconditioning; liver transplantation
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Intervention Model Description: Patients will be allocated to an intervention group (rIC) and compared to a retrospective control group. Data assessment will be blinded to the assessor.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patient enrolment will be done by the on-call doctor and intervention will be performed by unblinded research personnel who won't be involved in sample collection or data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (rIC) (Experimental): The rIC procedure will be applied on seated patients, who have been resting for at least five minutes. The active rIC procedure consists of four five-minute inflations of a pneumatic tourniquet to 100 mmHg above the patient's systolic blood pressure separated by five-minute periods of complete deflation. Placement of the pneumatic tourniquet will be unilaterally on a lower limb (right thigh)
  Interventions: Procedure: remote ischemic preconditioning (rIC)
- control group (non-rIC) (Other): The control group will be a retrospective group, who have undergone a liver transplantation and meet the inclusion criteria.
  Interventions: Other: non remote ischemic preconditioning (non-rIC)

INTERVENTIONS:
Procedure: remote ischemic preconditioning (rIC) — Short intermittent peripheral occlusions and reperfusions of the blood flow in the right lower extremity with the help of a tourniquet.
  Arms: intervention group (rIC)
Other: non remote ischemic preconditioning (non-rIC) — Retrospective group who have not undergone intervention.
  Arms: control group (non-rIC)

SUMMARY:
Ischemia and reperfusion injury is unavoidable during a liver transplantation. Remote ischemic preconditioning, a safe and feasible method, has previously been shown to reduce ischemia and reperfusion injury. In the transplantation setting, focus of remote ischemic preconditioning has been on the donor. However, preconditioning of the recipient may be a better approach due to the mechanisms by which ischemic preconditioning protects against ischemia and reperfusion injury.

The aim of this randomised, double-blinded clinical trial is to biochemically assess the liver function after application of remote ischemic preconditioning on the recipient.

DETAILED DESCRIPTION:
Background The use of solid organ transplantation, including liver transplantation, is the golden standard for many end-stage solid organ diseases. Ischemia and reperfusion injury is unavoidable during a liver transplantation. Remote ischemic preconditioning, a safe and feasible method, has previously been shown to reduce ischemia and reperfusion injury. This may have a similar effect in a liver transplantation setting. In the transplantation setting, focus of remote ischemic preconditioning has been on the donor. However, preconditioning of the recipient may be a better approach due to the mechanisms by which ischemic preconditioning protects against ischemia and reperfusion injury.

The aim of this randomised, double-blinded clinical trial is to biochemically assess the liver function after application of remote ischemic preconditioning on the recipient.

Methods 52 patients undergoing a liver transplantation, included in accordance to the inclusion criteria, will be allocated to an intervention group (rIC-group) and compared to a retrospective non-intervention control group (non-rIC group) consisting of 52 patients. Patients in the non-intervention group will also be included in accordance to the inclusion criteria. Within two hours before surgery, patients in the intervention group will be subjected to four rounds of five-minute inflations and five-minute deflations of a pneumatic tourniquet applied on the right leg.

Follow-up time will be 30 days.

Measurements The aim of this trial is to assess the effect of remote ischemic preconditioning on the extent of liver injury and inflammation as a result of ischemia and reperfusion injury. Assessment will be done by measurement of biomarkers relevant to liver function and liver injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver transplantation
* Patients aged 18 or above
* Patients who have given an informed consent

Exclusion Criteria:

* Patients undergoing re-transplantation.
* Patients who do not or cannot give an informed consent.
* Patients who have undergone surgery six weeks prior to liver transplantation.
* Patients with known peripheral vascular disease.
* Patients with an infection localized to the area of rIC-intervention
* Patients with at a high risk or with previous history of multiple thrombo-embolic diseases.
* Patients undergoing active immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Post-operative change in ALT | Day 0-4
  Extent of liver injury measured as change in ALT postoperative from day zero to day four .

SECONDARY OUTCOMES:
Post-operative change in Aspartate Amonitransferase | Day 0-4
  Serological markers of liver function
Post-operative change in Bilirubin | Day 0-4
  Serological markers of liver function
Post-operative change in Alkaline Phosphatase | Day 0-4
  Serological markers of liver function
Post-operative change in International Normalised Ratio | Day 0-4
  Serological markers of liver function

OTHER OUTCOMES:
Complication rate | Follow-up on day 30
  Rate of post-operative complications
Days in ICU (Intensive Care Unit) | Follow-up on day 30
  Length of post-operative stay in ICU
Total length of hospital-stay | Follow-up on day 30

CONTACTS AND LOCATIONS:
Overall Officials: Waqas Farooqui, MD, Principal Investigator — Doctor

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Farooqui W, Pommergaard HC, Rasmussen A. Remote ischemic preconditioning of transplant recipients to reduce graft ischemia and reperfusion injuries: A systematic review. Transplant Rev (Orlando). 2018 Jan;32(1):10-15. doi: 10.1016/j.trre.2017.06.001. Epub 2017 Jun 15. PMID 28637593